CLINICAL TRIAL: NCT02029690
Title: Phase 1 Study in Subjects With Tumors Requiring Arginine to Assess ADI-PEG 20 With Pemetrexed and Cisplatin (ADIPemCis) (TRAP Study)
Brief Title: Ph 1 Study in Subjects With Tumors Requiring Arginine to Assess ADI-PEG 20 With Pemetrexed and Cisplatin
Acronym: TRAP
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Polaris Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POLARIS2013-006
Record Dates: First submitted 2013-12-16; First posted 2014-01-08 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2019-03

CONDITIONS: Pleural Mesothelioma Malignant Advanced; Peritoneal Mesothelioma Malignant Advanced; Non-squamous Non-small Cell Lung Carcinoma; Uveal Melanoma; Hepatocellular Carcinoma; Glioma; Sarcomatoid Carcinoma
Keywords: argininosuccinate synthetase; arginine; arginine deiminase
MeSH Terms: conditions — Uveal Melanoma; Carcinoma, Hepatocellular; Glioma; Carcinoma | interventions — ADI PEG20

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADI-PEG 20 (Experimental): Arginine deiminase formulated with polyethylene glycol
  Interventions: Drug: ADI-PEG 20

INTERVENTIONS:
Drug: ADI-PEG 20

SUMMARY:
A study of ADI-PEG 20 (pegylated arginine deiminase), an arginine degrading enzyme in patients with histologically proven advanced malignant pleural mesothelioma (MPM), advanced peritoneal mesothelioma (in dose escalation cohort only), non-squamous non-small cell lung carcinoma stage IIIB/IV (NSCLC), metastatic uveal melanoma, hepatocellular carcinoma (HCC), glioma and sarcomatoid cancers

DETAILED DESCRIPTION:
Weekly ADI-PEG 20 will be cohort dose escalated (18, 27 and 36 mg/m2), with pemetrexed 500 mg/m2 and cisplatin 75 mg/m2 both given every 3 weeks. Subjects may receive a maximum of 6, 3-week cycles of ADIPemCis for a total of 18 weeks of treatment. Subjects with NSCLC may receive 4 to 6, 3-week cycles as per local institutional policy. Those subjects completing ADIPemCis treatment may continue on ADI-PEG 20 monotherapy if they have SD or better. Subjects with NSCLC may continue to receive pemetrexed as per local institutional policy along with ADI-PEG 20 and/or continue on ADI-PEG 20 monotherapy after pemetrexed is also discontinued.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven advanced MPM, advanced peritoneal mesothelioma (for dose escalation cohort only) or non-squamous NSCLC (stage IIIB/IV) who have not been treated with prior chemotherapy or immunotherapy, except that NSCLC subjects with EGFR mutant or ALK positive must have had an EGFR tyrosine kinase inhibitor (TKI) or ALK inhibitor and progressed or been shown to be intolerant of therapy prior to enrolling in this trial, if such ALK inhibitor and EGFR targeted therapy are approved and available in the country in which patients are being enrolled OR Histologically proven metastatic uveal melanoma who have not been treated with prior chemotherapy (MTD cohort only), OR Histologically proven HCC who have failed (PD and/or side effects-been intolerant of) treatment with sorafenib. Failure is defined as having progressed radiographically on, or been intolerant to prior systemic therapy. Intolerance is defined as discontinuation due to an AE(s) on prior systemic therapy that was unacceptable to the treating physician and / or patient, with or without dose interruption and modification. Failure requires at least 14 days of treatment with sorafenib, except for a subject that has had a severe allergic reaction to sorafenib at any time, even less than 14 days of treatment with sorafenib and thus it would be imprudent to re-challenge them with that agent. Cirrhotic status of Child-Pugh grade A-B7 must be present. Child-Pugh status should be determined based on clinical findings and laboratory data during the screening period (Appendix E). Subjects on anti-coagulants are to receive 1 point for their INR status, as they are presumed to have a <1.7 baseline PT/INR.", OR Histologically proven high-grade glioma who have failed (PD and/or side effects) treatment with radiotherapy ± temozolomide, OR Sarcomatoid cancer of any line.
2. ASS1 deficiency (defined as ≤50% ASS expression) demonstrated on tissue specimen (cytospin samples are acceptable) by immunohistochemistry (IHC). For subjects previously treated with chemotherapy, this specimen may have been obtained before that chemotherapy. A new tissue specimen obtained after most recent chemotherapy is not required. Thus ASS1 deficiency is required for entrance into the study. If tissue is not available to determine ASS1 deficiency, then tissue must be obtained by biopsy to determine ASS1 status.
3. Measurable disease as assessed by modified RECIST for MPM and by RECIST 1.1 criteria for peritoneal mesothelioma, NSCLC, uveal melanoma, HCC, glioma and sarcomatoid carcinoma
4. ECOG performance status of 0 - 1
5. Predicted life expectancy of at least 12 weeks.

Exclusion Criteria:

1. Radiotherapy (except for palliative reasons), targeted therapy, or immunotherapy (except for uveal melanoma) the previous four weeks before study treatment.
2. Ongoing toxic manifestations of previous treatments.
3. Symptomatic brain or spinal cord metastases (patients must be stable for > 3 months post radiotherapy or surgery) for subjects with mesothelioma, NSCLC, uveal melanoma excludes subjects with HCC or glioma).
4. Major thoracic or abdominal surgery from which the patient has not yet recovered.
5. Serious infection requiring treatment with intravenous antibiotics at the time of study entrance, or an infection requiring intravenous therapy within 7 days prior to the first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-04-23 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Define initial estimates of efficacy, measured by RECIST 1.1 criteria for non-squamous NSCLC, advanced peritoneal mesothelioma, metastatic uveal melanoma, HCC, glioma and sarcomatoid cancers for ADI-PEG 20 in combination with pemetrexed and cisplatin. | 18 weeks
Define initial estimates of efficacy, measured by modified RECIST criteria for advanced MPM | 18 weeks

SECONDARY OUTCOMES:
Determine the MTD of ADI-PEG 20 in combination with pemetrexed and cisplatin | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szlosarek, MD, PhD, Principal Investigator — Barts Cancer Institute
Locations (4):
- Mayo Clinic Rochester, Rochester, Minnesota, United States
- United Kingdom (3):
  - Centre for Experimental Cancer Medicine (CECM), London, England
  - Cambridge Hospital, Cambridge
  - Guys Hospital, London

REFERENCES:
- [Derived] Chan PY, Phillips MM, Ellis S, Johnston A, Feng X, Arora A, Hay G, Cohen VML, Sagoo MS, Bomalaski JS, Sheaff MT, Szlosarek PW. A Phase 1 study of ADI-PEG20 (pegargiminase) combined with cisplatin and pemetrexed in ASS1-negative metastatic uveal melanoma. Pigment Cell Melanoma Res. 2022 Jul;35(4):461-470. doi: 10.1111/pcmr.13042. Epub 2022 May 16. PMID 35466524
- [Derived] Szlosarek PW, Wimalasingham AG, Phillips MM, Hall PE, Chan PY, Conibear J, Lim L, Rashid S, Steele J, Wells P, Shiu CF, Kuo CL, Feng X, Johnston A, Bomalaski J, Ellis S, Grantham M, Sheaff M. Phase 1, pharmacogenomic, dose-expansion study of pegargiminase plus pemetrexed and cisplatin in patients with ASS1-deficient non-squamous non-small cell lung cancer. Cancer Med. 2021 Oct;10(19):6642-6652. doi: 10.1002/cam4.4196. Epub 2021 Aug 12. PMID 34382365
- [Derived] Hall PE, Lewis R, Syed N, Shaffer R, Evanson J, Ellis S, Williams M, Feng X, Johnston A, Thomson JA, Harris FP, Jena R, Matys T, Jefferies S, Smith K, Wu BW, Bomalaski JS, Crook T, O'Neill K, Paraskevopoulos D, Khadeir RS, Sheaff M, Pacey S, Plowman PN, Szlosarek PW. A Phase I Study of Pegylated Arginine Deiminase (Pegargiminase), Cisplatin, and Pemetrexed in Argininosuccinate Synthetase 1-Deficient Recurrent High-grade Glioma. Clin Cancer Res. 2019 May 1;25(9):2708-2716. doi: 10.1158/1078-0432.CCR-18-3729. Epub 2019 Feb 22. PMID 30796035